CLINICAL TRIAL: NCT00092833
Title: An Open-Label, Worldwide, Treatment Use Study to Provide Ezetimibe 10 Mg/Day to Patients With Homozygous Familial Hypercholesterolemia or Homozygous Sitosterolemia
Brief Title: Investigational Drug in Patients With Hypercholesterolemia or in Patients With Sitosterolemia (0653-026)(COMPLETED)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0653-026; 2004_034
Record Dates: First submitted 2004-09-23; First posted 2004-09-28 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia, Familial; Lipid Metabolism, Inborn Errors
MeSH Terms: conditions — Hyperlipoproteinemia Type II; Lipid Metabolism, Inborn Errors

ARMS (1):
- 1 (Experimental): Ezetimibe
  Interventions: Drug: Comparator: ezetimibe

INTERVENTIONS:
Drug: Comparator: ezetimibe — Ezetimibe (MK0653) 10 mg once daily for 3 years.

SUMMARY:
The purpose of this study is to provide an investigational drug to patients with a specific type of hypercholesterolemia (high cholesterol) or sitosterolemia (unusually high absorption of non-cholesterol sterols) in a treatment use setting.

ELIGIBILITY:
Inclusion Criteria:

* Homozygous familial hypercholesterolemia or sitosterolemia

Exclusion Criteria:

* Patient has a condition which, in the opinion of the investigator, might pose a risk to the patient, interfere with participation in the study, or does not meet the additional criteria as required by the study

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2002-07; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Incidence of clinical and laboratory adverse experiences in in patients with homozygous FH or homozygous sitosterolemia taking ezetimibe 10 mg/day | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC